CLINICAL TRIAL: NCT00656045
Title: The Effects of Two Different Leisure-time Activity Prescriptions on Eating and Activity Behaviors During Behavioral Weight Loss Treatment
Brief Title: Leisure Time Activity and Nutrition Program
Acronym: LEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEAN E01-1703-011
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Obesity; Physical Activity
Keywords: Obesity; Physical Activity; Weight Loss; Exercise; Dietary Intake; Energy; Behavioral; Healthy Eating
MeSH Terms: conditions — Obesity; Motor Activity; Weight Loss; Behavior | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Arm A focuses on increasing the participant's physical activity level.
  Interventions: Behavioral: Dietary; Behavioral: Physical Activity
- B (Experimental): Arm B focuses on decreasing the amount of time the participant spends watching Television.
  Interventions: Behavioral: Dietary; Behavioral: TV Watching

INTERVENTIONS:
Behavioral: Dietary — All participants in the investigation will receive a standard 8-week behavioral obesity intervention with 8 weekly, 1 hour group counseling and education sessions. The intervention will include a reduced caloric prescription (1200-1500 kcal/day) and fat gram prescription (30% or less kcals from fat).
Behavioral: Physical Activity — The Physical Activity arm will receive an activity goal (200 minutes/week of moderate-intense physical activity).
  Arms: A
Behavioral: TV Watching — The TV Watching arm will receive a TV watching goal of watching less than 10 hours of TV/week.
  Arms: B

SUMMARY:
The purpose of this investigation is to conduct an 8-week pilot study to examine the effects of two different leisure-time activity prescriptions on dietary intake, leisure-time activities, and weight loss in 26 adults receiving a standard 8-week behavioral weight loss intervention.

DETAILED DESCRIPTION:
In adult observational studies, TV viewing has been positively related to overweight and obesity. It is theorized that TV watching influences eating and activity behaviors, such that with greater TV watching less physical activity and greater consumption of energy occurs, producing a positive energy balance state. While no experimental research has been conducted with adults examining the influence of reducing TV watching on weight status, experimental research conducted with children does indicate that lower levels of TV watching can produce reduced energy intake and greater levels of physical activity. Most importantly, family-based, behavioral childhood obesity interventions that have targeted reducing sedentary behaviors (which includes TV watching) have found that as compared to targeting increasing physical activity during treatment, similar increases in activity and fitness occur, but that greater weight loss and greater increases in liking for physical activity occur when sedentary behaviors, as compared to physical activity, are targeted in family-based behavioral childhood weight control programs.

Thus, this investigation will involve an 8-week pilot study to examine the effects of two different leisure-time activity prescriptions. All participants in the investigation will receive a standard 8-week behavioral obesity intervention. The intervention will include a reduced caloric prescription (1200-1500 kcal/day) and fat gram prescription (30% or less kcals from fat). One condition will receive an activity goal (200 minutes/week of moderate-intense physical activity [Physical Activity]), while the other condition will receive a TV watching goal (10 hours/week [ TV Watching]). Participants will be assessed at 0 and 9 weeks (pre- and post-intervention) on measures of dietary intake, physical activity, TV watching, liking of physical activity and TV watching, and weight.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 and 40 kg/m2
* Watch > 16 hours per week of TV
* Engage in < 100 minutes of moderate-intense physical activity per week

Exclusion Criteria:

* Participants reporting a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q). Individuals self-reporting joint problems, prescription medication usage related to heart conditions, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
* Reporting they are unable to walk for 2 blocks (1/4 mile) without stopping.
* Reporting no TVs in the home or 5 or more TVs in the home viewed by the participant (TVs in participant's children's bedrooms will not be counted).
* Reporting major psychiatric diseases or organic brain syndromes via a phone screen.
* Participating in a weight loss program and/or taking weight loss medication or that have lost > 5% of body weight during the past 6 months.
* Participating in a program to increase physical activity and/or decrease TV watching time.
* Intending to move to another city within the time frame of the investigation.
* Being pregnant, lactating, less than 6 months post-partum, or planning to become pregnant during the time frame of the investigation.
* Having had gastric surgery for weight loss.
* Being unwilling to attend weekly sessions.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Time spent in moderate-intense physical activity | 8 weeks

SECONDARY OUTCOMES:
Weight loss | 8 weeks
Caloric and fat intake while watching TV | 8 weeks
Liking of physical activity | 8 weeks
Time spent watching TV | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A. Raynor, Ph.D., Principal Investigator — University of Tennessee; David Bassett Jr., Ph.D., Study Chair — University of Tennessee; Dixie Thompson, Ph.D., Study Chair — University of Tennessee; Amy Gorin, Ph.D., Study Chair — University of Connecticut
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States

REFERENCES:
- See also: This is the website for the Healthy Eating and Activity Laboratory (HEAL), where this program is being conducted. — http://heal.utk.edu/